CLINICAL TRIAL: NCT03466190
Title: Clinical Assessment of Postoperative Occlusion in Patient With Mandibular Body Fractures Reduced and Fixed With Computer-assisted Polyether Ether Ketone (PEEK) Custom Made Plates Versus Conventional Titanium Plates (RCT)
Brief Title: Clinical Assessment of Computer-assisted PEEK Versus Conventional Titanium Plates on Mandibular Body Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rofaida Atef Atef, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-02-27
Record Dates: First submitted 2018-03-02; First posted 2018-03-15 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Fracture Mandible; Mandibular Fractures
Keywords: Mandibular body fractures, PEEK plates, titanium plates.
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Intervention Model Description: * A Randomized clinical trial.
  * A trial will be carried out in hospital of Oral and Maxillofacial surgery department- Faculty of Oral and Dental Medicine Cairo University
  * Equal randomization: participants with equal probabilities for intervention.
  * Positive controlled: Both groups receiving treatment.
  * Parallel group study: Each group of patients receives a single treatment simultaneously.
Masking Description: Because the two interventions used in this trial are clearly different and easily recognized by the participants and investigators, neither the investigator nor participants can be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Custom made PEEK plate fixation (Experimental): Open Reduction Internal Fixation using Custom made PEEK plates.
  Interventions: Procedure: Custom made PEEK plate fixation
- Titanium plate fixation (Active Comparator): Open Reduction Internal Fixation using conventional titanium plating system.
  Interventions: Procedure: Titanium plate fixation

INTERVENTIONS:
Procedure: Titanium plate fixation — Under General Anesthesia, exposure of the fractured mandibular body segments will be done using a standardized surgical approach. Open Reduction Internal Fixation using conventional titanium plates will be performed.
  Other Names: Conventional titanium plates
  Arms: Titanium plate fixation
Procedure: Custom made PEEK plate fixation — Under General Anesthesia, exposure of the fractured mandibular body segments will be done using a standardized surgical approach. Open Reduction Internal Fixation using custom made PEEK plates will be performed.
  Other Names: Computer-assisted PEEK plate fixation
  Arms: Custom made PEEK plate fixation

SUMMARY:
Two groups of patients with mandibular body fractures indicated for Open reduction internal fixation alone or in combination with fractures elsewhere in the mandible or midface. First group will be subjected to traditional titanium internal rigid fixation. Second group will be subjected to custom made PEEK plates.

DETAILED DESCRIPTION:
Two groups of patients with mandibular body fractures indicated for Open reduction internal fixation alone or in combination with fractures elsewhere in the mandible or midface. First group will be subjected to traditional titanium internal rigid fixation. Second group will be subjected to custom made PEEK plates.

Inclusion criteria:

All subjects were required:

1. Patients with at least a unilateral body fracture indicated for Open reduction internal fixation alone or in combination with fracture elsewhere in the mandible or midface.
2. All ages and both sexes were included in this study.
3. Patients should be free from any systemic disease that may affect normal healing of bone, and predictable outcome.
4. Patients with good general condition allowing major surgical procedure under general anesthesia.
5. Patients with physical and psychological tolerance.

Exclusion criteria:

1. Patients with high risk systemic diseases like uncontrolled diabetes . As uncontrolled diabetes has a negative impact on normal bone healing.
2. Patients with old fractures. As they will affect accuracy of reduction of the fractured segments.
3. Patients with physical and psychological intolerance. As psychological stress will affect the immune system and patient's fitness including healing capacity.

Interventions:

Eligible patients will be randomized in equal proportions between the study group (PEEK custom made plates) and the control group (titanium plates).

A- Computer-assisted PEEK custom made plates:

* All cases will undergo surgery under general anesthesia.
* Exposure of the fractured segments will be done using a standardized surgical approach.
* The fractured segments will be reduced in normal anatomic position guided by customized plate.
* Fracture fragments will be fixed using PEEK custom made plate utilizing 2.0 mm screws.

B- Conventional titanium plates:

* All cases will undergo surgery under general anesthesia.
* Exposure of the fractured segments will be done using a standardized surgical approach.
* Inter-maxillary fixation will be done.
* The fractured segments will be reduced in normal anatomic position guided by occlusion.
* The fracture fragments will be fixed using 2.3 titanium plate on the inferior border and 2.0 titanium plate on the superior border utilizing bone screws.

Follow up:

Clinical evaluation will be performed at the first week postoperative. Computed tomography will be performed at the first week postoperative then patients will be recalled for clinical evaluation every week for one month. Final follow up visit will be at 3 months postoperative.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with at least a unilateral body fracture indicated for Open reduction internal fixation alone or in combination with fracture elsewhere in the mandible or midface.
2. All ages and both sexes were included in this study.
3. Patients should be free from any systemic disease that may affect normal healing of bone, and predictable outcome.
4. Patients with good general condition allowing major surgical procedure under general anesthesia.
5. Patients with physical and psychological tolerance.

Exclusion Criteria:

1. Patients with physical and psychological intolerance. Because psychological stress will affect the immune system and general health.
2. Patients with systemic diseases like uncontrolled diabetes mellitus. Because uncontrolled diabetes mellitus has a negative impact on normal bone healing.
3. Patients with old and/or mal-union fractures. As they will affect accuracy of reduction of the fractured segments.
4. Patient with bad oral hygiene. As it has an influence on normal osseous healing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-08-02 (Actual); Primary Completion 2019-03-02 (Estimated); Study Completion 2019-03-02 (Estimated)

PRIMARY OUTCOMES:
Postoperative occlusion | 1 month postoperative
  Restoration of normal patient occlusion will be assessed using Visual analog scale (VAS)
  (0-10)

SECONDARY OUTCOMES:
Accuracy of the planned reduction | 1st week
  The accuracy of computer assisted PEEK custom made plates in open reduction and
  internal fixation of mandibular body fractures will be assessed using Mimics software, measuring unit (mm)
Wound dehiscence | 1 month postoperative
  Wound infection will be assessed via clinical assessment, measuring unit (Binary yes/no)
The need for 2nd surgery | 1 month postoperative
  Redo surgery will be assessed via clinical assessment, measuring unit (Binary yes/no)
Operative time | During operation
  Surgical time will be assessed via clinical assessment, measuring unit (hours)

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Amr, PhD, Study Director — Faculty of Oral and Dental Medicine -Cairo University
Locations (1):
- Faculty of Oral and Dental Medicine -Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Open reduction and rigid internal fixation of mandibular condylar fractures by an intraoral approach: a long-term follow-up study of 15 patients — http://www.ncbi.nlm.nih.gov/pubmed/17113444
- See also: Accuracy of the Computer-Aided Surgical Simulation (CASS) System in the Treatment of Patients With Complex Craniomaxillofacial Deformity: A Pilot Study. — https://www.ncbi.nlm.nih.gov/pubmed/?term=Accuracy+of+the+Computer-Aided+Surgical+Simulation+(CASS)+System+in+the+Treatment+of+Patients+With+Complex+Craniomaxillofacial+Deformity%3A+A+Pilot+Study.
- See also: A Comparative Evaluation of Fixation Techniques in Anterior Mandibular Fractures Using 2.0 mm Monocortical Titanium Miniplates Versus 2.4 mm Cortical Titanium Lag Screws — http://link.springer.com/10.1007/s12663-012-0342-1
- See also: Titanium osteosynthesis hardware in maxillofacial trauma surgery: to remove or remain? A retrospective study. — https://www.ncbi.nlm.nih.gov/pubmed/26814516
- See also: Camerani, et al. Reconstruction of frontal bone using specific implant polyether-ether-ketone — http://www.ncbi.nlm.nih.gov/pubmed/22075823
- See also: The effect of diabetes mellitus on osseous healing. — https://www.ncbi.nlm.nih.gov/pubmed/20465554
- See also: Unfavourable outcomes in maxillofacial injuries: How to avoid and manage — http://www.ncbi.nlm.nih.gov/pubmed/24501458
- See also: Stress-induced immune dysregulation: Implications for wound healing, infectious disease and cancer — https://www.ncbi.nlm.nih.gov/pubmed/18040814